CLINICAL TRIAL: NCT00178620
Title: PATCAR Pilot Trial: A Phase 4 Study, Pre-hospital Administration of Thrombolytic Therapy With Urgent Culprit Artery Revascularization
Brief Title: Pre-hospital Administration of Thrombolytic Therapy With Urgent Culprit Artery Revascularization
Acronym: PATCAR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Richard Smalling, Professor - Internal Medicine, Cardiology, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PATCAR Pilot Trial HSC 03-021
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Results first posted 2023-09-06 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Heart Disease; Myocardial Infarction; Acute Myocardial Infarction
Keywords: Heart Disease; Heart Attack; Myocardial Infarction; Thrombolytic Therapy; Emergency Medicine
MeSH Terms: conditions — Heart Diseases; Myocardial Infarction | interventions — reteplase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group A: Full dose pre-hospital fibrinolysis (Experimental): Patients transported by participating EMS units and that were fibrinolytic eligible and treated with full dose, pre-hospital fibrinolysis with reteplase (treated in the ambulance with 10 units reteplase and randomized to a second 10-unit dose of reteplase).
  Interventions: Drug: Reteplase 10 Units (U) plus a second dose of reteplase 10 U
- Group B: Half dose pre-hospital fibrinolysis followed by urgent PCI (Experimental): Patients transported by participating EMS units and that were fibrinolytic eligible and treated with a half dose pre-hospital fibrinolysis with reteplase (treated in the ambulance with 10 units reteplase) and randomized to urgent catheterization with percutaneous coronary intervention (PCI).
  Interventions: Drug: Reteplase 10 U; Procedure: Urgent Percutaneous Coronary Intervention (PCI)
- Group C: Fibrinolytic ineligible patients receiving primary PCI (Active Comparator): Patients transported by participating EMS units and that were fibrinolytic ineligible and treated with primary PCI alone and that were prospectively analyzed for comparison.
  Interventions: Procedure: Primary Percutaneous Coronary Intervention (PCI)
- Group D: Patients transferred in and treated with primary PCI (Active Comparator): Patients not transported by participating EMS units but were transferred in and treated with primary PCI alone and that were prospectively analyzed for comparison.
  Interventions: Procedure: Primary Percutaneous Coronary Intervention (PCI)

INTERVENTIONS:
Drug: Reteplase 10 Units (U) plus a second dose of reteplase 10 U — Thrombolytic-clot busting drug Retavase IV Bolus, 10 U followed by a second 10U dose
  Other Names: Retavase
  Arms: Group A: Full dose pre-hospital fibrinolysis
Drug: Reteplase 10 U — Thrombolytic-clot busting drug Retavase IV Bolus in one 10U dose
  Other Names: Retavase
  Arms: Group B: Half dose pre-hospital fibrinolysis followed by urgent PCI
Procedure: Urgent Percutaneous Coronary Intervention (PCI)
  Arms: Group B: Half dose pre-hospital fibrinolysis followed by urgent PCI
Procedure: Primary Percutaneous Coronary Intervention (PCI)
  Arms: Group C: Fibrinolytic ineligible patients receiving primary PCI; Group D: Patients transferred in and treated with primary PCI

SUMMARY:
The PATCAR study has been designed to test the hypothesis that the strategy of pre-hospital use of a "clot busting" (thrombolytic) drug followed with emergent heart catheterization including stenting of the problematic coronary artery, will result in a lower mortality and reduced repeat heart attack rates.

Early identifying and treating heart attacks patients prior to the arriving at the hospital, in those patients who qualify for the "clot busting" drugs will lower the size of the heart attack damage. This smaller heart attack will lead to fewer problems with less repeat heart attacks and death in the future.

DETAILED DESCRIPTION:
To demonstrate feasibility of the project in a pilot trial we plan to enroll up to 500 patients to pre-hospital thrombolysis/clot busting followed by emergent catheterization and stenting of the problematic or culprit artery.

This will comprise an EMS system capable of performing pre-hospital ECGs followed by emergent transportation to a Level I Cardiovascular Center where the patients will be taken to urgent cardiac catheterization and emergent stenting of the culprit artery.

Patients identified as having typical symptoms of acute MI and an ECG consistent with acute ST elevation MI will be screened in the field by paramedics or in the spoke hospitals by the ED attending physicians using the screening form. Verbal Consent will be obtained for receiving acute therapy for their MI as outlined in the protocol. After therapy is initiated in the field or at the spoke hospital, the patients will be transported as quickly as possible to the receiving Level I Cardiovascular Center (Hub Hospital). The ED personnel in the Level I Cardiovascular Center will have activated the Interventional Cardiovascular Team and the Cath Lab personnel after having received the initial qualifying transmitted ECG.

Once the patient arrives, informed consent will be obtained by the ED investigator and/or in-house Cardiology fellow for enrollment in the PATCAR Trial. Thrombolytic ineligible patients will also be collect for this study and also go directly to the Cath Lab for PCI. Study coordinators will enter the data into the Case Report Forms and forward the completed forms to Westat-ALA for data capture in the database. In addition to the qualifying ECG, ECG's will be obtained at hospital discharge/transfer. All patients will follow the current standard of care for STEMI/heart attacks patients. Patients will have a Cardiac MRI done on day 3 or 5 of their hospital stay, to measure the size and amount of damage the heart suffered as a result of their Heart attack.

ELIGIBILITY:
Inclusion Criteria:

1. Ischemic discomfort (squeezing, crushing, or pressure, sub-sternal, unrelated to breathing or movement), epigastric discomfort or pre-syncopal symptoms with diaphoresis, lasting > 30 minutes.
2. ST elevation > 0.1 mV in 2 or more contiguous limb leads or > 0.2 mV in 2 or more contiguous pre-cordial leads.
3. Less than 6 hours after onset of sustained chest pain.
4. Age 18 years or older.

Exclusion Criteria:

1. Chest pain described as ripping or tearing, radiating to the back and/or down the leg, and/or systolic blood pressure > 15 mmHg difference in each arm.
2. Suspected cocaine or amphetamine use within previous 3 days.
3. Known or suspected pregnancy.
4. Cardiac arrest requiring intubation.
5. Cardiac arrest requiring greater than 20 minutes CPR.
6. Coronary intervention (PTCA/stent/CABG) within previous 4 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Actual)
Dates: Start 2003-09 (Actual); Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard W. Smalling, MD, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Memorial Hermann Hospital / The University of Texas HSC, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All ACS patients 18 years or older with documented STEMI on EKG, who presented within 6 hours of onset of sustained chest pain, and met all eligibility criteria, were enrolled in PATCAR after an informed consent was obtained.
Groups:
- Group A: Full dose, pre-hospital fibrinolysis followed by treatment in the coronary care unit
- Group B: One-half dose pre-hospital reteplase followed by urgent PCI
- Group C: Fibrinolytic ineligible patients, treated with primary PCI at the STEMI center
- Group D: Patients not transported by participating EMS units but were transferred in and treated with primary PCI at the STEMI center
Period: Overall Study
Arm/Group | Group A | Group B | Group C | Group D
Started | 37 | 253 | 37 | 63
Completed | 37 | 253 | 37 | 63
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group C: Fibrinolytic ineligible patients who were treated with primary PCI at the STEMI center.
- Group D: Patients not transported by participating EMS units transferred in and treated with primary PCI at the STEMI center.
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Group D | Total
Number analyzed (Participants) | 37 | 253 | 37 | 63 | 390
Age, Customized [Number; unit: participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 37 | 253 | 37 | 63 | 390
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 69 | 17 | 14 | 106
  Male | 31 | 184 | 20 | 49 | 284
Treatment Allocation by Group [Number; unit: participants] | 37 | 253 | 37 | 63 | 390

OUTCOME MEASURES:

1. Primary Outcome: Mortality at 30 Days
Time Frame: 30 day
Measure: Number; unit: participants
Groups:
- Group A: Full does, pre-hospital fibrinolysis followed by treatment in the coronary care unit.
Arm/Group | Group A | Group B | Group C | Group D
Number analyzed (Participants) | 37 | 253 | 37 | 63
participants | 1 | 7 | 3 | 2

2. Secondary Outcome: Infarction Size as Measured by Cardiac Magnetic Resonance Imaging (MRI)
Time Frame: 1 year
Population: Data were not collected for this outcome measure.
Arm/Group | Group A | Group B | Group C | Group D
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Reduction in Time From Onset of Pain to Reperfusion
Time Frame: 1 year
Population: Data were not collected for this outcome measure.
Arm/Group | Group A | Group B | Group C | Group D
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Angiographic Documentation of Reperfusion
Time Frame: 1 year
Population: Data were not collected for this outcome measure.
Arm/Group | Group A | Group B | Group C | Group D
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Electrocardiogram (ECG) ST Segment Elevation Recovery
Time Frame: 1 year
Population: Data were not collected for this outcome measure.
Arm/Group | Group A | Group B | Group C | Group D
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Group A | Group B | Group C | Group D
Serious Adverse Events (participants affected / at risk) | 0/37 | 9/253 | 4/37 | 0/63
Other Adverse Events (participants affected / at risk) | 0/37 | 0/253 | 0/37 | 0/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=37) | Group B (N=253) | Group C (N=37) | Group D (N=63)
Death (Cardiac disorders) | 0 (0) | 9 (9) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No